CLINICAL TRIAL: NCT03261232
Title: Prognostic Factors in Refractory Cardiac Arrest Treated With Extracorporeal Life Support at Dijon CHU
Brief Title: Search for Prognostic Factors Associated With Better Survival in Refractory Cardiac Arrest
Acronym: Pro-ACR
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: ELLOUZE 2016 Pro-ACR
Record Dates: First submitted 2017-08-23; First posted 2017-08-24 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Cardiac Arrest (CA); ExtraCorporeal Life Support (ECLS)
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Through this retrospective observational study (over 4 years; period analysed: 1st January 2011 to 31st December 2014), we looked for prognostic factors associated with better survival in refractory cardiac arrest by:

* assessing the overall survival rate
* evaluating the frequency of intra et extra-hospital events and by comparing these with the survival rate
* studying no flow, low flow, rhythm at initial management, troponinemia, lactatemia and blood pH in the different groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with in-hospital or out-of-hospital refractory CA who underwent ECLS

Exclusion Criteria:

* CA occurring during cardiac surgery
* Age > 75 years or < 18 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with in-hospital or out-of-hospital refractory CA who underwent ECLS
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Survival rate | at baseline
Death rate | at baseline

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Ellouze O, Vuillet M, Perrot J, Grosjean S, Missaoui A, Aho S, Malapert G, Bouhemad B, Bouchot O, Girard C. Comparable Outcome of Out-of-Hospital Cardiac Arrest and In-Hospital Cardiac Arrest Treated With Extracorporeal Life Support. Artif Organs. 2018 Jan;42(1):15-21. doi: 10.1111/aor.12992. Epub 2017 Sep 6. PMID 28877346